CLINICAL TRIAL: NCT00099047
Title: Biologic and Clinical Role of COX-2 Inhibitor (Celecoxib)in the Management of MGUS and Smoldering Myeloma
Brief Title: Celecoxib in Preventing Multiple Myeloma in Patients With Monoclonal Gammopathy or Smoldering Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2009-00866; NCI-2009-00866 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000393514; UARK-18697; MAYO-206904; CCF-IRB-7029 (Other: Cleveland Clinic Foundation); N01-CN-25140 (Other: DCP); N01CN25140 (Other: US NIH Grant/Contract Award Number)
Record Dates: First submitted 2004-12-08; First posted 2004-12-09 (Estimated); Results first posted 2015-06-09 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Monoclonal Gammopathy of Undetermined Significance; Multiple Myeloma; Smoldering Multiple Myeloma
MeSH Terms: conditions — Monoclonal Gammopathy of Undetermined Significance; Multiple Myeloma; Smoldering Multiple Myeloma | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (celecoxib) (Experimental): Patients receive celecoxib PO BID for 6 months in the absence of unacceptable toxicity or progression to malignancy.
  Interventions: Drug: celecoxib; Other: laboratory biomarker analysis
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO BID for 6 months in the absence of unacceptable toxicity or progression to malignancy.
  Interventions: Drug: placebo; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: celecoxib — Given PO
  Other Names: Celebrex
  Arms: Arm I (celecoxib)
Drug: placebo — Given PO
  Arms: Arm II (placebo)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial studies how well celecoxib works in preventing multiple myeloma in patients with monoclonal gammopathy or smoldering myeloma. Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. The use of celecoxib may be effective in preventing multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OJBECTIVES:

I. Determine the efficacy of celecoxib vs placebo in reducing serum levels of M-component in patients with monoclonal gammopathy of undetermined significance or smoldering myeloma.

SECONDARY OBJECTIVES:

I. Determine the effects of this drug on secondary biomarkers as surrogate endpoints in these patients.

OUTLINE:

This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to participating center and type of monoclonal gammopathy (monoclonal gammopathy of undetermined significance vs smoldering myeloma). Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive celecoxib orally (PO) twice daily (BID) for 6 months in the absence of unacceptable toxicity or progression to malignancy.

ARM II: Patients receive placebo PO BID for 6 months in the absence of unacceptable toxicity or progression to malignancy.

After completion of study treatment, patients are followed at 1, 6, and 12 months.

ELIGIBILITY:
Criteria:

* M-protein >= 30 g/L
* No clinical evidence of chronic infectious or inflammatory disease
* No present evidence of active malignancy (nonmelanoma skin cancer or cervical intraepithelial neoplasia allowed)
* No hypersensitivity (e.g., asthma, urticaria, or acute rhinitis induced by NSAIDs) to aspirin or other NSAIDs
* No hypersensitivity to sulfonamides
* No uncontrolled diabetes
* No history of diabetic retinopathy
* No condition that would preclude study participation
* No condition that would preclude the use of NSAIDs
* New or preexisting diagnosis of 1 of the following for at least 2 months:
* Monoclonal gammopathy of undetermined significance as defined by the following criteria:
* M-protein =< 30 g/L
* Bone marrow clonal plasma cells < 10% and low level of plasma cell infiltration in a trephine biopsy (if done)
* Smoldering myeloma as defined by at least 1 of the following criteria:
* Bone marrow clonal plasma cells >= 10%
* No related organ or tissue impairment (i.e., end organ damage) or symptoms
* Asymptomatic patients with =< 3 lytic lesions (without other organ damage) attributable to plasma cell dyscrasia allowed
* No condition associated with a secondary monoclonal gammopathy
* IgG, IgA, or light chain M-component >= 1.0 g/dL for at least 2 consecutive lab readings taken at least 4 weeks apart
* No anemia
* No hepatic insufficiency
* AST or ALT < 1.5 times upper limit of normal (ULN)
* Bilirubin =< 1.5 times ULN
* Creatinine =< 1.8 mg/dL
* No hypercalcemia
* No renal insufficiency
* No uncontrolled congestive heart failure
* No history of cerebrovascular or cardiovascular accident
* No history of gastrointestinal hemorrhage
* No active or suspected peptic ulcer disease
* Previously treated H. pylori infection allowed
* More than 12 months since limited chemotherapy
* More than 28 days since prior chronic or frequent use of glucocorticoids (> 5 mg of prednisone or equivalent per day)
* More than 28 days since prior chronic or frequent use of non-steroidal anti-inflammatory drugs (NSAIDs) (> 100 mg of aspirin per day)
* More than 28 days since prior bisphosphonate therapy
* More than 28 days since prior investigational agents
* Concurrent low-dose aspirin ( =< 100 mg/day) allowed
* No evidence of other B-cell proliferative disorders (e.g., multiple myeloma, Waldenstrom's macroglobulinemia, primary amyloidosis, or lymphoproliferative disease)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* AND/OR
* ECOG 0-1 or Zubrod 0-1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2004-11; Primary Completion 2008-06 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matt Kalaycio, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 23 asymptomatic adult patients with a serum monoclonal protein >1g/dL from Cleveland Clinic, Mayo Clinic, or University of Arkansas Medical Center were randomized between August 2005 and April 2008
Pre-assignment Details: There were no significant events or approaches utilized following enrollment but prior to group assignment.
Period: Overall Study
Arm/Group | Arm I (Celecoxib) | Arm II (Placebo)
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Asymptomatic adult patients with a serum monoclonal protein >1g/dL from each of the participating centers between August 2005 and April 2008 were randomized to either celecoxib or placebo in a double-blind, 1:1 fashion
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Celecoxib) | Arm II (Placebo) | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 17
  >=65 years | 3 | 3 | 6
Gender [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 6 | 8 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 10 | 12 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 11 | 11 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 12 | 23
serum monoclonal protein >1g/dL [Number; unit: participants] | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Changes in M-protein Levels
Description: For a given biomarker (or a suitable transformation of it, e.g. log transform) t-tests and Wilcoxon tests (2-sample t-test and Wilcoxon rank sum test for between treatment comparisons, and paired 1-sample t-test and Wilcoxon signed rank test for within treatment comparisons) will be used to detect statistically significant differences between (or within) treatments.
Time Frame: Baseline and 6 months
Population: One patient on the celecoxib arm was considered inevaluable and not included in this participants analyzed.
Measure: Median (Standard Deviation); unit: g/dL
Arm/Group | Arm I (Celecoxib) | Arm II (Placebo)
Number analyzed (Participants) | 10 | 12
g/dL | 1.65 (0.36) | 2.24 (0.36)
Statistical Analysis 1: Comparison: Arm I (Celecoxib) vs Arm II (Placebo); Test type: Superiority or Other; p = .23, SAS version 8; Median Difference (Final Values) = .05, Standard Deviation .05 — 36 evaluable patients randomized 1:1 to each treatment was planned in order to have >77% power to detect differences in above parameters equal to or greater than one standard deviation, based on a 2-sided Wilcoxon rank-sum test with .05 Type I error

ADVERSE EVENTS:
Arm/Group | Arm I (Celecoxib) | Arm II (Placebo)
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 6/11 | 8/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Celecoxib) (N=11) | Arm II (Placebo) (N=12)
headache (Nervous system disorders) | 2 (2) | 4 (4)
Fatigue (General disorders) | 1 (1) | 2 (2)
Pruritus/Itching (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Neuorpathy (Nervous system disorders) | 2 (2) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Exremity Limb Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (5)
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain NOS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Upper Respiratory (Infections and infestations) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
No overall limitations or caveats for this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less